CLINICAL TRIAL: NCT04877925
Title: Coaxial Drainage Versus Standard Chest Tube After Pulmonary Lobectomy: a Randomized Controlled Study
Brief Title: Coaxial Drainage Versus Standard Chest Tube After Pulmonary Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Anile (Other)
Responsible Party: Sponsor-Investigator, Marco Anile, Principal Investigator, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COAXIAL
Record Dates: First submitted 2021-04-27; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Group (Active Comparator): Patients with 2 standard chest tubes
  Interventions: Device: standard chest tubes
- Coaxial Group (Experimental): Patients with 1 coaxial tube
  Interventions: Device: coaxial chest tube

INTERVENTIONS:
Device: standard chest tubes — 2 standard postoperative chest tube used
  Arms: Standard Group
Device: coaxial chest tube — 1 postoperative smart drain coaxial tube
  Arms: Coaxial Group

SUMMARY:
Objectives: Chest tubes are routinely inserted after thoracic surgery procedures in different size and numbers. The aim of this study is to assess the efficacy of Smart Drain Coaxial drainage compared with two standard chest tubes in patients undergoing thoracotomy for pulmonary lobectomy. 98 patients (57 males and 41 females, mean age 68.3±7.4 years) with lung cancer undergoing open pulmonary lobectomy were randomized in two groups: 50 received one upper 28-Fr and one lower 32-Fr standard chest tube (ST group) and 48 received one 28-Fr Smart Drain Coaxial tube (CT group). Hospitalization data, quantity of fluid output, air leaks, radiograph findings, pain control and costs were assessed.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years
* patients scheduled for pulmonary lobectomy

Exclusion Criteria:

* middle lobectomy,
* extended resections, minimally invasive lobectomies,
* previous ipsilateral thoracic surgery,
* induction chemo and/or radiotherapy
* patients who did not give consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Daily fluid drainage (mL) | 1 postoperative day
  Quality of fluid drainage evaluated in mL and by means of a chest X rays
Presence of postoperative pneumothorax | 1 postoperative day
  Quality of air drainage evaluated by chest X rays

SECONDARY OUTCOMES:
presence of pneumothorax after tubes removal | within 24 hours after tubes removal
  Pneumothorax evaluated by chest x rays
evaluation of pain measured by Visual Analogue Scale | 1 postoperative day
  evaluation of patient's pain with a 1 - 10 scale ( 0 no pain - 10 maximum pain)
Analysis of costs (in euros) | until discharge, an average of 6 days
  Evaluation of hospital costs in euros during the hospitalization
Postoperative hospitalization (in days) | until discharge, an average of 6 days
  Duration of hospitalization in days after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guerrera F, Filosso PL, Pompili C, Olivetti S, Roffinella M, Imperatori A, Brunelli A. Application of the coaxial smart drain in patients with a large air leak following anatomic lung resection: a prospective multicenter phase II analysis of efficacy and safety. J Vis Surg. 2018 Jan 29;4:26. doi: 10.21037/jovs.2018.01.07. eCollection 2018. PMID 29445612
- [Result] Rena O, Parini S, Papalia E, Massera F, Turello D, Baietto G, Casadio C. The Redax(R) Coaxial Drain in pulmonary lobectomy: a study of efficacy. J Thorac Dis. 2017 Sep;9(9):3215-3221. doi: 10.21037/jtd.2017.08.110. PMID 29221298